CLINICAL TRIAL: NCT06152094
Title: UCSF BP Activate Letter Randomized Clinical Trial
Brief Title: UCSF BP Activate Letter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37619
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BP Activate Letter (Experimental): Participants in the BP Activate Letter arm will receive a BP Report letter that includes computerized algorithm recommendations for medication changes they should discuss with their clinician.
  Interventions: Other: BP Activate Letter
- Control Letter (Active Comparator): Participants in the Control Letter arm will receive a Control letter suggesting they talk to their clinician about their blood pressure (without BP history or specific medication recommendations).
  Interventions: Other: Control Letter
- Usual Care (No Intervention): Participants in the Usual Care arm will not receive any letter or any other intervention.

INTERVENTIONS:
Other: BP Activate Letter — Participants in the BP Activate Letter arm will receive a BP Activate Report that includes personalized details about recent measurements, current medications, and "computer-generated medication recommendations that might improve your blood pressure", along with a log for tracking additional SMBP measurements. They will also receive a cover letter that includes an assessment that BP appears to be uncontrolled, and suggesting a visit with their provider to discuss.
  Arms: BP Activate Letter
Other: Control Letter — Participants in the Control Letter arm will receive a cover letter that includes an assessment that BP appears to be uncontrolled, and suggesting a visit with their provider to discuss.
  Arms: Control Letter

SUMMARY:
The BP Activate Study aims to assess the effectiveness of the BP Report letter with personalized BP medication recommendations, compared with Control letters and no intervention, at shortening time to appointment, time to visit, time to medication change, and time to achievement of BP goal.

DETAILED DESCRIPTION:
The BP Activate Study is a randomized quality improvement trial. We will deliver one of two versions of a letter to established English-speaking primary care patients at Mt Zion with uncontrolled hypertension, defined by SBP>140 or DBP>90 in the past two years (identified via EHR). The letter will prompt patients to schedule a visit with their provider or team nurse practitioner to discuss their BP recommendations with their clinician. We will test 2 versions of the letter and a usual care control:

1. The "BP Activate Report Letter" group will get a letter that presents recommendations for medication changes from a computerized algorithm using the patient's medical records and recommends discussing these specific recommendations with their clinician; or
2. The "Control Letter" group will get a letter that suggests they talk to their clinician about their BP without providing any specific medication recommendations.
3. The "Usual Care" group will not receive any intervention.

This primary goal of the study is to assess the effectiveness of the BP Activate Report Letter compared with the Control Letter, and see if it shortens time to appointment, time to visit, time to medication change (primary outcome), and time to achievement of BP goal. Clinicians, with patient input, will still have full control of how BP is clinically managed. A small number of patients will be contacted by a research coordinator to hear what they thought when they received the letter, and why they did or did not act upon the information.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a primary care patient of a clinician in a general internal medicine clinic who has agreed to have their patients participate in the study
* Lowest SBP>140 or lowest DBP>90 at last visit in general internal medicine clinic
* Last visit in general internal medicine clinic was < 2 years ago
* EngageRx algorithm determines that a medication intensification step is indicated

Exclusion Criteria:

* Primary language is not English
* Patient's provider indicates (through an active opt-out process) that they do not want the patient to receive a BP Activate letter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time to medication change or demonstrated BP control at 6 months | 6 months
  Time is measured as number of days between randomization date and the day that a participant is prescribed a new anti-HTN medication or an increase in dose of a prior anti-HTN medication, or they have a documented BP measurement <140 mmHg systolic and <90 mmHg diastolic.

SECONDARY OUTCOMES:
Time to medication change or demonstrated BP control at 3 months | 3 months
  Time is measured as number of days between randomization date and the day that a participant is prescribed a new anti-HTN medication or an increase in dose of a prior anti-HTN medication, or they have a documented BP measurement <140 mmHg systolic and <90 mmHg diastolic.
Time to completed visit at 3 months | 3 months
  Time to medication change is defined as number of days between randomization and the day the participant completes a visit in the Division of General Internal Medicine.
Time to BP goal at 3 months | 3 months
  Time is defined as number of days from randomization until first documentation of a BP measurement <140 mmHg systolic and <90 mmHg diastolic.
Time to medication change at 3 months | 3 months
  Time is measured as number of days between randomization date and the day that a participant is prescribed a new anti-HTN medication or an increase in dose of a prior anti-HTN medication.
Time to completed visit at 6 months | 6 months
  Time to medication change is defined as number of days between randomization and the day the participant completes a visit in the Division of General Internal Medicine.
Time to BP goal at 6 months | 6 months
  Time is defined as number of days from randomization until first documentation of a BP measurement <140 mmHg systolic and <90 mmHg diastolic.
Time to medication change at 6 months | 6 months
  Time is measured as number of days between randomization date and the day that a participant is prescribed a new anti-HTN medication or an increase in dose of a prior anti-HTN medication.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pletcher, MD MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No